

### STATISTICAL ANALYSIS PLAN

A Phase IIb, Randomized,

Double Blind, Placebo Controlled Dose Ranging Study to

Assess the Effect of RPL554 in Patients with Moderate to

Severe COPD

**Study No. RPL554-CO-203 Version 1.0 – 6 March 2018** 



### Statistical Analysis Plan

Verona Pharma RPL554-CO-203

### **Authorization Signature Page**

A Phase IIb, Randomized, Double Blind, Placebo Controlled Dose Ranging Study to Assess the Effect of RPL554 in Patients with Moderate to Severe COPD

Eleonora Chiossi Statistical Scientist

IQVIA

Author:

Approved by:

Mark Shaw

Associate Director, Biostatistics

**IQVIA** 

**Customer Representative:** 

Kenneth Newman, MD, MBA

Chief Medical Officer

Verona Pharma Plc



### **Modification History**

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 1.0 | 6 March 2018 | Eleonora Chiossi | Final Version for implementation after DB lock |



### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation or special term | Explanation/Definition |
|---|---|
| AEs | Adverse Events |
| ANCOVA | Analysis of Covariance |
| ATS | American Thoracic Society |
| AUC | Area under the curve |
| BDI | Baseline Dyspnea Index |
| BID | Twice a day |
| BMI | Body Mass Index |
| Bpm | Beats per Minute |
| CIs | Confidence Intervals |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRF | Case Report Form |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| E-RS | Evaluating – Respiratory Symptoms |
| ERS | European Respiratory Society |
| EXACT-PRO | Exacerbations of Chronic Pulmonary Disease Tool Patient-Reported Outcome |
| $FEV_1$ | Forced expiratory volume in 1 second |
| FVC | Forced Vital Capacity |
| ICS | Inhaled corticosteroids |
| Kg | Kilograms |
| LABA | Long Acting Beta <sub>2</sub> Agonist |
| LAMA | Long Acting Muscarinic Antagonist |
| LDL | Low-density Lipoprotein |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| m | Meters |
| mL | Milliliters |
| MMRM | Mixed Model for Repeated Measures |
| MRC | Medical Research Council |
| msec | Milliseconds |
| N | Number of patients |
| PGAC | Patient Global Assessment of Change |
| PT | Preferred Term |
| QTcF | QT interval corrected for heart rate using Friderica's formula |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SGRQ-C | St George's Respiratory Questionnaire – COPD specific |
| TDI | Transition Dyspnea Index |



### **Table of Content**

| 1. | Intro | ductionduction | 7 |
|---|---|---|---|
| 2. | Study | objectives | 7 |
| | 2.1. | Primary objective | 7 |
| | 2.2. | Secondary objectives | 7 |
| | 2.3. | Exploratory Objectives | 7 |
| 3. | Study | design | 8 |
| | 3.1. | General Description | |
| | 3.2. | Treatments | 8 |
| | | 3.2.1. Treatments Administered | 8 |
| | | 3.2.2. Method of Assigning Patients to Treatment Groups | |
| | | 3.2.3. Blinding | |
| | 3.3. | Determination of Sample Size | |
| | 3.4. | Changes in the Conduct of the Study or Planned Analyses | |
| | 3.5. | Analysis Sets | 9 |
| | 3.6. | Major Protocol Deviations | 10 |
| | 3.7. | General Methodology | 10 |
| | | 3.7.1. Baseline | |
| | | 3.7.2. End of Study | |
| | | 3.7.3. Visit Windows | |
| | | 3.7.5. Treatment period. | |
| | 3.8. | Handling of Dropouts or Missing Data | |
| | | 3.8.1. Missing data in efficacy analysis | 11 |
| | | 3.8.2. Missing data in safety analysis | |
| | | 3.8.3. Partial Date Imputation | |
| | | 3.8.4. Partial Dates for AEs | |
| | 3.9. | Interim Analyses and Data Monitoring | |
| | 3.10. | Pooled country/region | |
| 4 | | | |
| 4. | | nt disposition, demographic and baseline characteristics, medical his and concomitant medications, treatment compliance and exposure | |
| | 4.1. | Patient disposition | |
| | 4.2. | Demographic and Other Baseline Characteristics | |
| | 4.3. | Medical History | |
| | 4.4. | Prior COPD, Prior and Concomitant Medications | |
| | | 4.4.1. Special grouping of medications. | |
| | 4.5. | Exposure and compliance | |
| | - | 4.5.1. Treatment Compliance | |
| | | 4.5.2. Extent of Exposure | 15 |
| 5. | Effica | acy Endpoints | 15 |





| | 5.1. | Primary Efficacy Endpoint | 15 |
|---|---|---|---|
| | 5.2. | Secondary Efficacy Endpoints | 16 |
| | 5.3. | Exploratory Efficacy Endpoints | 16 |
| | 5.4. | Selected secondary endpoints | 17 |
| | 5.5. | Efficacy Endpoints details | 17 |
| | | 5.5.1. Pulmonary Function Tests | |
| | | 5.5.2. Symptom Diary [EXACT-PRO] | |
| | | 5.5.3. St. George's Respiratory Questionnaire – COPD specific (SGRQ-C) | |
| | | 5.5.4. Medical Research Council (MRC) Breathlessness Scale | |
| | | 5.5.5. Patient Global Assessment of Change (PGAC) | |
| | <i>5.6</i> | 5.5.6. Baseline and Transition Dyspnea Indices (BDI and TDI) | |
| | 5.6. | Efficacy Endpoint Analysis | |
| | | <ul><li>5.6.1. General consideration on the analysis of efficacy</li><li>5.6.2. Analysis of Primary Endpoint</li></ul> | |
| | | 5.6.3. Analyses of Secondary and exploratory Endpoints | |
| | | 5.6.4. Multiple Comparison Adjustment for the Primary Efficacy Endpoint | |
| | | 5.6.5. Multiple Comparison Adjustment for the Secondary Efficacy Endpoint | |
| | | 5.6.6. Examination of Subgroups | |
| 6. | Safet | y Endpoints | 22 |
| | 6.1. | Adverse Events | 22 |
| | | 6.1.1. Analysis of Adverse Events | 22 |
| | 6.2. | Clinical Laboratory Evaluations | |
| | | 6.2.1. Analysis of Clinical Laboratory Evaluation | |
| | 6.3. | Electrocardiograms | |
| | | 6.3.1. Analysis of ECG Evaluations | 24 |
| | | 6.3.2. Holter Monitors | 24 |
| | 6.4. | Vital Signs | 24 |
| | | 6.4.1. Analysis of Vital Signs | 25 |
| | 6.5. | Physical Findings | 25 |
| | 6.6. | Drug induced bronchospasm | 25 |
| | | 6.6.1. Analysis of drug induced bronchospasm | 25 |
| 7. | Phar | macokinetic | 25 |
| | 7.1. | Analysis of pharmacokinetic | 25 |
| 8. | REFI | ERENCES | 27 |
| 9. | | endices | |
| ۶. | 9.1. | Appendix 1: Schedule of Events | |
| | 9.2. | Appendix 2: EXACT-PRO Scoring Instructions | |
| | 9.3. | Appendix 3: SGRQ-C | |
| | 9.4 | Appendix 4: SAS code for efficacy analysis | 38 |


Version: 1.0 Version Date: 6 March 2018



### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for protocol RPL554-CO-203. It describes, in detail, the data to be summarized and analyzed, including specifics of the statistical analyses to be performed. This statistical analysis plan is based on the final protocol version 2.0, dated 18<sup>th</sup> of April 2017.

### 2. Study objectives

The purpose of this study is to investigate the dose response of RPL554 in patients with Chronic Obstructive Pulmonary Disease (COPD) over 4 weeks. Clinical practice indicates that this length of time should allow for the study of the bronchodilator response (measured predominantly by peak FEV<sub>1</sub>) and the anti-inflammatory response (measured predominantly by trough FEV<sub>1</sub>).

### 2.1. Primary objective

The primary objective of this study is to investigate the placebo-corrected effect of RPL554 administered by nebulizer on change from baseline in peak FEV1 (maximum over 3 hours following dosing) over 4 weeks when administered to patients with moderate to severe COPD.

### 2.2. Secondary objectives

The secondary objectives of this study are as follows:

- To investigate the placebo-corrected effect of RPL554 administered by nebulizer on change from baseline in morning trough FEV<sub>1</sub> over 4 weeks when administered to patients with moderate to severe COPD
- To investigate the bronchodilator placebo-corrected effect of RPL554 administered by nebulizer on AUC<sub>0-12</sub> hours FEV<sub>1</sub> after 4 weeks of dosing
- To investigate the single-dose bronchodilator placebo-corrected effect of RPL554 on peak and average FEV<sub>1</sub> at Visit 2 (first dose)
- To investigate the bronchodilator placebo-corrected effect of RPL554 on peak and average FEV<sub>1</sub> over 3 hours at Visits 3 to- 6 (Weeks 1 to 4)
- To investigate the placebo-corrected effects of RPL554 on COPD symptoms, as measured by daily diary (E-RS from the Exacerbations of Chronic Pulmonary Disease Tool Patient-Reported Outcomes [EXACT-PRO+], Transition Dyspnea Index [TDI], St George's Respiratory Questionnaire COPD specific [SGRQ-C], Medical Research Council [MRC] scale, and patient global assessment of change (PGAC)
- To investigate the safety of RPL554 when administered for 4 weeks in patients with COPD, as measured by adverse events, electrocardiograms (ECGs), Holter monitoring and vital signs
- To compare the amount of rescue albuterol/salbutamol use required

### 2.3. Exploratory Objectives

Additional, exploratory objectives of this study are as follows:

- To compare peak and AUC<sub>0-12 hour</sub> FEV<sub>1</sub> at the final study visit (visit 6) to baseline (Day 1)
- To correlate trough pharmacokinetics with pharmacodynamics effects

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx
Author: Eleonora Chiossi Version: 1.0
 Version Date: 6 March 2018



### 3. Study design

This is a phase IIb, randomized, double-blind, placebo-controlled, parallel group study designed to evaluate the efficacy and safety of nebulized RPL554 in patients with moderate to severe COPD over 4 weeks.

### 3.1. General Description

A total of approximately 400 patients between the ages of 40 and 75 years, inclusive, with a clinical diagnosis of COPD, as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines and symptoms compatible with COPD for at least 1 year prior to screening will be enrolled.

Patients will be seen at approximately 50 sites throughout the European Union. The study comprises six visits: screening (visit 1), randomization (visit 2), and weekly visits for 4 weeks (visit 3 to visit 6, Week 1 to Week 4). Patients will be screened for eligibility (visit 1), including a reversibility test with albuterol/salbutamol between 7 and 14 days before the first dose of study medication.

### 3.2. Treatments

### 3.2.1. Treatments Administered

Patients will be randomized to either RPL554 or placebo. Those assigned to RPL554 will receive one of four active strengths, as described in the table below:

| Substance | Dose Level (mg) | Concentration (mg/mL) |
|----------------------|-----------------|-----------------------|
| RPL554 | 0.75 | 0.3 |
| RPL554 | 1.5 | 0.6 |
| RPL554 | 3.0 | 1.2 |
| RPL554 | 6.0 | 2.4 |
| Placebo | N/A | N/A |
| N/A = Not Applicable | | |

**Table 1: RPL554 Doses** 

All study medications will be administered twice daily, using a standard jet nebulizer.

### 3.2.2. Method of Assigning Patients to Treatment Groups

At the screening visit, the investigator will assign a unique patient number to each enrolled patient. This patient number is made up of three digits unique to each study site and 3 digits for each consecutively enrolled patient at the trial site, provided an informed consent form is signed by the patient. This number should be entered into the electronic data capture (EDC) system and maintained throughout the study. Once the patient meets inclusion and exclusion criteria, the study site will request the study medication assignment using the Interactive Response System (IXRS).

### 3.2.3. Blinding

This is a randomized, double-blind, placebo-controlled study. Placebo will be similar to




RPL554, except for the omission of the active ingredient. Because a visually matching placebo could not be developed, the dosing cup on each nebulizer administered at the study center will be obscured with opaque tape to visually blind the study medication.

### 3.3. Determination of Sample Size

The standard deviation for peak FEV1 is estimated to be 250 mL. With a 2-sided test at a 5% significance level and 80 evaluable patients per group, there will be an 80% power to detect a true difference of 111 mL between any two treatments. This detectable limit has been considered sufficient to conclusively identify a minimal effective dose of RPL554. Thus 80 patients per group will be randomized for a total of 400 patients.

### 3.4. Changes in the Conduct of the Study or Planned Analyses

- The method for analysis the primary efficacy endpoint has been changed from LOCF ANCOVA to mixed model for repeated measures (MMRM). The change was led by the superiority of MMRM with respect to LOCF in avoiding some type of bias as suggested by Siddiqui et al. (Siddiqui O, 2009)
- Introduction of Per Protocol analysis set. This is an analysis set of interest for a phase II study.

### 3.5. Analysis Sets

All randomized analysis Set: includes all randomized patients

**Safety Analysis Set**: includes all patients who receive at least one dose of investigational product during the study. It is a subset of all randomized analysis set.

**Full Analysis Set**: includes all randomized patients, who receive at least one dose of investigational product during the study and with at least one post/treatment efficacy data assessment among spirometry EXACT-PRO questionnaire, SGRQ, TDI PGAC and MRC. It is a subset of the safety analysis set.

**Per-Protocol Analysis Set**: includes all patients who do not have pre-specified major protocol deviations which can affect the efficacy outcome or the treatment of the subject (see section 3.6). It is a subset of the safety analysis set.

Use of the analysis set

| | All- | Full Analysis | Safety | Per-Protocol |
|---|---|---|---|---|
| | Randomized | Set | Analysis Set | Analysis Set |
| | set | | | |
| Disposition of patients | X | | | |
| Protocol deviations | X | | | |
| Demographic and other | X | | | |
| baseline characteristics | | | | |
| Medical history | X | | | |
| Prior and concomitant | | | X | |
| medication | | | | |
| Treatment compliance and | | | X | |
| extent of exposure | | | | |

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx




| Efficacy: Primary endpoint | X | | X |
|----------------------------|---|---|---|
| Efficacy: Secondary | X | | X |
| endpoints | | | |
| Efficacy: Exploratory | X | | X |
| endpoints | | | |
| Safety | | X | |
| Pharmacokinetic | | X | |

The number and percentage of patients within each of these analysis sets will be presented by treatment group and overall.

### 3.6. Major Protocol Deviations

Major protocol deviations will be defined in a separate document that will be finalized before database lock.

Patients with major protocol deviations will be identified by a clinical review of the data prior to database lock to the extent possible in light of restrictions due to blinding of study personnel to treatment assignments.

A summary of major protocol deviations will be presented by treatment group for all randomized patients.

### 3.7. General Methodology

Summary statistics will be presented to give descriptions of patients and an overview of efficacy and safety results. All analysis tables will include summaries for all five treatment groups: RPL554 0.75 mg BID, RPL554 1.5 mg BID, RPL554 3.0 mg BID, RPL554 6.0 mg BID, Placebo BID. Categorical parameters will be summarized with number of observations and percentage of patients in each category. Continuous parameters will be summarized using number of observations, mean, standard deviation (SD), median, minimum and maximum.

Unless specified otherwise, all statistical tests will be two-sided. All p-values will be rounded to three decimal places; p-values less than 0.001 will be presented as '<0.001' and greater than 0.999 will be presented as '>0.999' in all tables.

All available data from all patients will be listed.

### 3.7.1. Baseline

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to study medication start date (including unscheduled assessments). In the case where the last non-missing measurement and the study medication start date coincide (and time is either not collected or missing), that measurement will be considered pre-baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

### 3.7.2. End of Study

This will be visit 6

### 3.7.3. Visit Windows

No visit windows will be applied in this study and the scheduled assessments will be reported and analyzed as per CRF collection.




### 3.7.4. Duration

For the purposes of calculating durations expressed in months, a month will be considered as one-twelfth of a year, or 365.25 / 12 = 30.4375 days.

As for duration in days, the calculation will go as follows:

- (stop date start date) + 1 if start date is same as first dose date or later;
- (stop date start date) if start date is before first dose date.

### 3.7.5. Treatment period

Treatment period is defined as the time elapsed between the first and last dose intake date plus 1 day. Assessments will be included in the safety and efficacy analysis if performed during the treatment period.

### 3.8. Handling of Dropouts or Missing Data

### 3.8.1. Missing data in efficacy analysis

MMRM model will be used as a strategy to deal with missing data.

Last observation carried forward approach (LOCF) will be used a sensitivity analysis of the primary endpoint only.

No other imputation will be applied.

### 3.8.2. Missing data in safety analysis

Any missing safety parameter will be considered missing for purposes of any summary statistics and analysis.

### 3.8.3. Partial Date Imputation

Dates are essential for the classification of AEs as treatment-emergent and medications as having been taken prior to the start of study medication and/or concomitantly with study medication.

### 3.8.4. Partial Dates for AEs

Adverse event start date (references to month are the month of the AE start date):

- 1. If only month and year are known and study medication started during that month then set start date equal to study medication start date.
- 2. If month and year are known and study medication started prior to or after that month then set start date equal to 1st day of month.
- 3. If only year is known, and it is the same as study medication start year, assume it is the study medication start date/year. If it is different from study medication start year, assume it is the first day of the year.
- 4. If full start date (i.e. day, month, and year are missing) is unknown impute start date as the study medication start date. If imputed start date is greater than stop date, it will be imputed as stop date.




### 3.8.5. Partial Dates for Concomitant Medications

Concomitant therapy start date (references to month are the month of the concomitant therapy start date). Partial date imputation will follow the same pattern as for AEs in section 3.8.4 above.

Concomitant therapy stop date (references to month are the month of the concomitant therapy stop date):

- 1. If only day is unknown, then set equal to last day of month.
- 2. If only year is known, assume it is the last day of the year.
- 3. Otherwise (i.e. day, month and year are missing) leave as missing.

### 3.9. Interim Analyses and Data Monitoring

There are no planned interim analyses of data from this study.

### 3.10. Pooled country/region

For all analyses, sites will be pooled within countries. This will be detailed and approved prior to database lock.

4. Patient disposition, demographic and baseline characteristics, medical history, prior and concomitant medications, treatment compliance and exposure

### 4.1. Patient disposition

The final patient disposition will be presented by treatment group and overall. The total number of patients randomized, treated, completed and discontinued (including reason for discontinuation as recorded on the CRF) from the study will be summarized by treatment group and overall. The total number of patients prematurely discontinued will be presented overall and by visit. If the patient has discontinued between Visit 2 and Visit 3 it will be counted on those discontinued up to Week 1, and so on.

### 4.2. Demographic and Other Baseline Characteristics

Demographics including age, age group, gender, ethnicity and race will be presented by treatment group and overall. Also, presented by treatment group and overall are the following baseline characteristics: post-bronchodilator FEV1 (both in liters and in percentage of predicted normal), post-bronchodilator FVC, FEV1/FVC, FEV1 reversibility test results, duration of COPD (from diagnosis to randomization), smoking habits.

Statistical testing will not be performed on these parameters.

### 4.3. Medical History

The number and percentage of patients in the SAF with at least one medical condition, diagnosis or surgery will be presented by treatment group and overall. Furthermore, the incidence for each System Organ Class (SOC) and Preferred Term (PT) will be presented. For each patient, multiple events that map to a SOC and PT will be counted only once for incidence counts. Events will be in descending frequency of SOC and PT in summaries. A listing of all medical history will also be presented.

Document: U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx




### 4.4. Prior COPD, Prior and Concomitant Medications

Prior medications are defined as medications taken prior to first study medication dose. Concomitant medications are defined as medications with onset dates on or after the first dose of study medication, or medications with onset dates prior to first dose of study medication without a stop date or with a stop date after first dose of study medication. Partial date imputation for medications is described in section 3.8.5.

Prior and concomitant medications will be classified by WHO Drug Dictionary that identifies the active ingredient.

Prior and concomitant medications will be summarized by therapeutic subgroup (ATC level 2), active ingredient and treatment group (for prior COPD medications and prior medications the overall column will also be presented), displaying frequencies and percentages. The denominators for the percentages will be the numbers of patients in each treatment group. Medications will be sorted by decreasing order of frequency of the therapeutic subgroup and active ingredient within subgroup.

A separate summary of patient taking COPD medications prior to the study by therapeutic class will also be presented. COPD medications are identified as those with 'Indication='COPD' on the medication log.

### 4.4.1. Special grouping of medications

Special grouping of beta agonist will be done as follows and will replace the ATC2 code classification.

### LAMAs

ATC4=R03BB and active ingredient equal to

- o tiotropium
- o umeclidinium
- o aclidinium

ATC4=A03AB and active ingredient equal

- o glycopyrronium
- LABAs

ATC4=R03AC and active ingredient equal to

- o salmeterol
- o formoterol
- indacaterol
- o olodaterol

ATC4=R03AK and active ingredient equal to

vilanterol and fluticasone furoate

ATC4=R03AL3 and active ingredient equal to

o vilanterol and umeclidinium bromide




### o vilanterol, umeclidinium bromide and fluticasone furoate

### • Inhaled corticosteroids (ICS)

ATC4 = R03BA or

ATC4= R03AK and active ingredient equal

- beclometasone
- budesonide
- o flunisolide
- betamethasone
- o fluticasone
- o triamcinolone
- o mometasone
- o ciclesonide
- o fluticasone furoate

### • LABA/LAMA

Active ingredient includes

- o 'glycopyrronium' and 'indacaterol'
- o 'olodaterol' and 'tiotropium'
- o 'aclidinium' and 'formoterol'
- o 'umeclidinium' and 'vilanterol'

### LABA/ICS

Active ingredient includes

- o 'budesonide' and 'formoterol'
- o 'fluticasone' and 'salmeterol'
- o 'fluticasone' and 'vilanterol'
- o 'beclomethasone' and 'formoterol'
- o 'mometasone' and 'formoterol'




### 4.5. Exposure and compliance

### 4.5.1. Treatment Compliance

Treatment compliance will be summarized by treatment group in 2 ways:

- 1. 100\*((number of vials dispensed number of vials returned)/(expected number of vials to be taken during study period)) (excluding visit 6 for completers, as the vials will be dispensed by the site)
- 2. Drug intake as recorded in the e-diary: percent of 'yes' responses. The denominator is the number of records for which the patient provided an answer (Yes or No) to drug intake questions (morning and evening) in the e-diary.

### 4.5.2. Extent of Exposure

Duration of exposure to study medication will be calculated as follows:

(Stop date - start date) + 1.

The mean duration of exposure in days will be summarized by treatment group. Total exposure (in mL) will be based on the number of vials dispensed against the number returned (number of vials\* contents of each vial (in mL)).

For in-clinic dosing, the RPL554 exposure will be calculated based on the nominal dose.

### 5. Efficacy Endpoints

### 5.1. Primary Efficacy Endpoint

- Change from baseline FEV<sub>1</sub> to peak FEV<sub>1</sub> (over 3 hours) at Week 4
  - o Baseline is defined as the FEV<sub>1</sub> pre-dose assessment (-15 minutes) collected at Visit 2
  - Peak FEV<sub>1</sub> at Week 4 is defined as the maximum post-dose value among the 30 minutes, 1, 2 and 3 hour assessments collected at Visit 6 (Week 4).

### **5.2.** Secondary Efficacy Endpoints

- Change from baseline FEV<sub>1</sub> to morning trough FEV<sub>1</sub> at Week 1, 2, 3 and 4
- Change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> (over 12 hours) at Day 1 and at Week 4
- Change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> (over 3 hours) at Day 1, Week 1, 2, 3, and
- Change from baseline FEV<sub>1</sub> to peak FEV<sub>1</sub> (over 3 hours) at Day 1, Week 1, 2 and 3

For details on the derivation of the above FEV<sub>1</sub>endpoints refer to section 5.5.1

- Change from baseline in EXACT-PRO E-RS score at Week 4
- Change from baseline in EXACT-PRO Total score at Week 4
- Change from baseline in EXACT-PRO E-RS Breathlessness score at Week 4
- Change from baseline in EXACT-PRO E-RS Cough/Sputum score at Week 4
- Change from baseline in EXACT-PRO E-RS Chest Symptoms score at Week 4



For details on the derivation of the above EXACT-PRO scores refer to section 5.5.2

- Change from baseline in the SGRQ-C Total score at Week 4
- Change from baseline in the SGRQ-C Symptoms score at Week 4
- Change from baseline in the SGRQ-C Activity score at Week 4
- Change from baseline in the SGRQ-C Impact score at Week 4

For details on the derivation of the above SGRQ-C scores refer to section 5.5.3

• Change from baseline in MRC breathlessness scales at Week 4

For details on the MRC scale refer to section 5.5.4

- Transition Dyspnea Index (TDI) at week 4
- Patient Global Assessment of Change (PGAC) at Week 4
- Change from baseline (average over the last 7 days of the run-in period) in average daily use of rescue medication over the treatment period, and at Week 1, 2, 3 and 4. Average daily use of rescue medication is the average of the number of times the rescue medications is taken (multiplied by two as two puffs are taken at each administration) during the period of time.

### 5.3. Exploratory Efficacy Endpoints

- Change from baseline in EXACT-PRO E-RS score at Week 1, 2 and 3
- Change from baseline in EXACT-PRO Total score at Week 1, 2 and 3
- Change from baseline in EXACT-PRO E-RS Breathlessness score at Week 1,2 and 3
- Change from baseline in EXACT-PRO E-RS Cough/Sputum score at Week 1,2 and 3
- Change from baseline in EXACT-PRO E-RS Chest Symptoms score at Week 1,2 and 3

For details on the derivation of the above EXACT-PRO scores refer to section 5.5.2

- Change from baseline in the SGRQ-C Total score at Week 2
- Change from baseline in the SGRQ-C Symptoms score at Week 2
- Change from baseline in the SGRQ-C Activity score at Week 2
- Change from baseline in the SGRQ-C Impact score at Week 2

For details on the derivation of the above SGRQ-C scores refer to section 5.5.3

• Change from baseline in MRC breathlessness scales at Week 2

For details on the MRC scale refer to section 5.5.4

- Transition Dyspnea Index at week 2
- Patient Global Assessment of Change (PGAC) at Week 2
- COPD exacerbation
  - O Patient with one adverse event with MedDRA Preferred Term='COPD exacerbation' and use of systemic steroids (ATC2=H02) from AE date of onset for at least three days
- Change in peak FEV<sub>1</sub> (over 12 hours) from Day 1 (single dose) to Week 4 (steady state)

### **5.4.** Selected secondary endpoints

The following secondary endpoints are of particular clinical interest and will undergo further




sensitivity analyses like subgroup analyses.

- Change from baseline FEV<sub>1</sub> to peak FEV<sub>1</sub> (over 3 hours) at Week 4
- Change from baseline FEV<sub>1</sub> to morning trough FEV<sub>1</sub> at Week 4
- Change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> (over 12 hours) at Week 4

### 5.5. Efficacy Endpoints details

### 5.5.1. Pulmonary Function Tests

<u>Baseline FEV<sub>1</sub></u> is defined as the FEV<sub>1</sub> pre-dose assessment (-15 minutes) collected at Visit 2.

<u>Peak FEV1 (over 3 (12) hours)</u> is defined as the maximum post-dose value among the values collected up to 3 (12) hours.

Morning trough FEV<sub>1</sub> is defined as the last pre-dose value at the visit under analysis

<u>Average FEV<sub>1</sub> (over 3 (12) hours)</u> is defined as the Area under the curve AUC<sub>0-3</sub> (AUC<sub>0-12</sub>) of the FEV1 values collected during the visit under analysis, divided by the length of the time (in hours) interval of interest. The AUC is calculated using the trapezoidal rule.

Parameters will be calculated over 3 hours (at Day 1 and Week 1 to 4) and over 12 hours (Day 1 and Week 4).

If patient miss hour 2 and 3 then the AUC 0-3 is set to missing. If patient miss hour 8 and 12 then AUC 0-12 is set to missing.

**Censoring of value after rescue medications:** before derivation of endpoints, within each visit, the spirometry data collected after the use of rescue medications (either Albuterol / Salbutamol or Ipratropium as collected on the CRF) will be censored (i.e.: considered as missing)

### **5.5.2.** Symptom Diary [EXACT-PRO]

Once patients provide answers to all 14 questions on the ePRO, the device produces a score for each of three subscales: breathlessness, cough/sputum and chest symptoms. In addition to the subscale scores, a total score (covering all 14 questions) and a score for the E-RS part (11 questions) together with the subscores will be obtained.

The average over the week 1, 2, 3 and 4 will be used as timepoint values, while the one over the week just prior to randomization (visit 2) will be used as baseline. If less than 4 days are available, the average over that week is set to missing.

Scoring will be performed as described in Appendix 2: EXACT-PRO and E-RS Scoring Instructions .

Note that, as the data are collected with an e-diary, there is no possibility of having missing items in the questionnaire as the system does not allow the patient to skip items. Also note that the EXACT-PRO subscale scores are not endpoints of the study but will be summarized for eventual comparison with other published studies

### 5.5.3. St. George's Respiratory Questionnaire – COPD specific (SGRQ-C)

Patients will be asked to complete the SGRQ-C while they are at the study site at Visits 2




(baseline), 4 and 6. This is a 14-question, multiple-choice questionnaire that has 2 parts. Part 1 (questions 1-7) produces the <u>symptoms score</u>, while part 2 (questions 8-14) produces the <u>activity</u> and <u>impacts</u> scores. A <u>total score</u> is also produced. Each possible answer to each of the 14 questions is assigned a weigh as in Appendix 3: SGRQ-C (Jones P. , 2012). The lowest possible weight is zero, the highest is 100. A single response is required to each item. With electronic collection, it is impossible that there could be multiple responses given to any one item.

The SGRQ-C is scored in 2 steps:

1. Sum the weights for all items with a positive response

The **<u>symptoms component</u>** score is obtained by adding the weights for items 1 through 7.

The <u>activity component</u> score is obtained by adding the weights for the positive responses to items Questions 9 and 12.

The <u>impacts component</u> score is obtained by adding the weights of items 8, 10, 11, 13 and 14 in the following way: the weights for all positive responses to items in Questions 10, 11 and 13 are summed together with the response to the single item that should have been checked/ticked in Questions 8 and 14.

### 2. Calculate the score

The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the result as a percentage.

$$Score = 100* \frac{Summed\ weights\ from\ all\ positive\ items\ in\ that\ component}{sum\ of\ maximum\ weights\ for\ all\ items\ in\ that\ component}$$

The total score is calculated similarly

$$Score = 100* \frac{Summed\ weights\ from\ all\ positive\ items\ in\ the\ questionnaire}{sum\ of\ maximum\ weights\ for\ all\ items\ in\ the\ questionaire}$$

The total score is calculated by summing the weights to all the positive responses in each component.

Please note that by "positive items", it is meant those that show the presence of symptoms, to some degree. For example, in question 1 (part 1), all answers ("most days", "several days" and "with chest infections") except "not at all" would be positive. Another way to identify a positive response from a negative one is that a positive response has a nonzero score, unlike a negative one. The same definition is true in part 2. With question 8 for example ("How would you describe your chest condition"?), the following responses are positive: "the most important problem I have", "causes me a few problems"; an answer of "Causes no problem" would be deemed negative as it does not show any signs of symptoms. In question 14 (see Appendix 3: SGRQ-C), as another example, any answer except "It does not stop me doing anything I would like to do" would be considered positive.

Note that, as the data are collected with an e-diary, there is no possibility of having missing items in the questionnaire as the system does not allow the patient to skip items.



### 5.5.4. Medical Research Council (MRC) Breathlessness Scale

The MRC is the most commonly used, validated scale to assess dyspnea in daily living in chronic respiratory diseases (Mahler & Wells, 1988) (Hajiro, et al., 1998). During Visits 2 (baseline), 4 and 6, patients will be provided with

the MRC (shown in Table 2 below) and asked on a grade of 1 to 5 how they would describe their levels of breathlessness.

 Grade
 Degree of breathlessness related to activities

 1
 Not troubled by breathlessness except on strenuous exercise

 2
 Short of breath when hurrying on the level or walking up a slight hill

 3
 Walks slower than most people on the level, stops after a mile or so, or stops after 15 minutes walking at own pace

 4
 Stops for breath after walking about 100 yds or after a few minutes on level ground

 5
 Too breathless to leave the house, or breathless when undressing

**Table 2: MRC Breathlessness Scale** 

This scale will be summarized at the time points at which it is collected, which are the same as SGRQ-C.

### 5.5.5. Patient Global Assessment of Change (PGAC)

At visits 4 and 6, patients will be asked to respond to a PGAC question along the following lines: "compared with prior to the study start, how do you feel your breathing is?" Answers are expected to use a 1-5 scale, where 1=much worse to 5=much better, with 3= no change. Answers will be summarized at visits 4 and 6, when the questionnaire is administered.

### 5.5.6. Baseline and Transition Dyspnea Indices (BDI and TDI)

The BDI and TDI are interviewer-administered ratings of dyspnea severity. They are based on three components that evoke dyspnea in activities of daily living. The questionnaires are comprised of 24 items covering 3 domains.

The domains are the following:

• For BDI: Functional impairment, magnitude of task and magnitude of effort. Patients are asked to recall during the previous 2 weeks. Each of these components ranges from 0 to 4

The BDI Total Score is the sum of the three domains and can take values from 0 to 12 (12 meaning no dyspnea) and is only assessed at baseline. The lower the score, the worse the dyspnea severity.

• For TDI: Change in functional impairment, change in magnitude of task, change in magnitude of effort. Each of these components ranges from -3 (major deterioration) to +3 (major improvement)

The TDI assesses the patient perception of the change in dyspnea severity from baseline. The TDI total score is the sum of the three TDI domains and can take values from -9 to 9. As with the BDI, the lower the TDI score, the more severe the dyspnea.

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx



### 5.6. Efficacy Endpoint Analysis

### **5.6.1.** General consideration on the analysis of efficacy

All efficacy analyses will be performed on the Full Analysis Set. Patients will be analyzed according to the randomized treatment. All efficacy summaries will present the five treatment groups. All data summarized will also be listed.

### 5.6.2. Analysis of Primary Endpoint

The primary efficacy analysis parameter is change from baseline  $FEV_1$  to peak  $FEV_1$  at Week 4 of treatment. The primary analysis will be based on the full analysis set.

Summary statistics for FEV<sub>1</sub> will be presented for baseline, week 4 and change from baseline by treatment group on patients with both assessments.

The primary analysis will use a restricted maximum likelihood (REML)—based repeated-measures approach. The change from baseline FEV<sub>1</sub> (at Day 1, Week 1, 2 3 and 4) will be the dependent variable. The analyses will include the fixed, categorical effects of treatment, visit, and treatment-by-visit interaction as well as the continuous, fixed covariates of baseline value. An unstructured (co)variance structure shared across treatment groups will be used to model the within-patient errors. If the model does not converge a compound symmetry (co)variance structure will be used. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom and adjust standard errors. Analyses will be implemented with SAS PROC MIXED (see Appendix 4: SAS code for efficacy analysis). The primary comparison will be the contrast (difference in least squares mean [LSMEAN]) between treatments at Week 4.

### 5.6.2.1. Sensitivity analysis for the primary endpoint

To check the robustness of the results the following analysis will be performed:

- MMRM analysis excluding the patients with only one on treatment assessment of peak FEV1 (over 3 hours)
- analysis of covariance (ANCOVA) will be used on data where missing data will be imputed using last observation carried forward (LOCF) method.

### 5.6.3. Analyses of Secondary and exploratory Endpoints

The secondary and exploratory endpoints will be analyzed in the same way as the primary endpoint.

In the analysis of TDI, BDI scores will be used as baseline in the model and the dependent endpoint will be the TDI score.

As for PGAC the model will not include the baseline as the score reflect itself a change from baseline.

The number of COPD exacerbations and use of rescue medications will be summarized by counts and percentages.

### 5.6.4. Multiple Comparison Adjustment for the Primary Efficacy Endpoint

The MMRM model above will test for the significance of treatment effect. Testing will continue



with each of the 4 doses of RPL554 against placebo, starting with the highest dose (6 mg).

To this end, the fixed-sequence testing approach (Maurer et al., 1995; (Westfall & Krishen, 2001)) will be used.

Let i = 0, 1, ..., 4 represent increasing dose levels, 0 denoting placebo. Also, let  $\mu_i$ , i = 0, 1, ..., 4, denote the mean change from baseline in peak FEV<sub>1</sub> after 4 weeks of treatment for placebo and each increasing active dose level, respectively. The primary null hypotheses are defined as:  $H_i$ :  $\mu_i - \mu_0 = 0$  and will be tested against the two-sided alternative  $K_i$ :  $\mu_i - \mu_0 \neq 0$ , i = 1, ..., 4.

Finally, let  $p_1, ..., p_4$  denote the marginal p-values obtained from the statistical tests associated with  $H_1, ..., H_4$  (obtained from the MMRM model).

The fixed-sequence testing will begin with the null hypothesis corresponding to the highest dose versus placebo. If a statistically significant difference is found at the two-sided  $\alpha$  level of 5%, the testing will proceed with the next highest dose, and so on. Otherwise, testing stops and the remaining null hypotheses are accepted without testing.

This testing strategy can be written as the following stepwise algorithm:

- Step 1: If  $p_4 \le \alpha$  reject  $H_4$  and go to Step 2. Otherwise accept  $H_1, ..., H_4$  and stop.
- Step 2: If  $p_3 \le \alpha$  reject  $H_3$  and go to Step 3. Otherwise accept  $H_1, ..., H_3$  and stop.
- Step 3: If  $p_2 \le \alpha$  reject  $H_2$  and go to Step 4. Otherwise accept  $H_1$  and  $H_2$  and stop.
- Step 4: If  $p_1 \le \alpha$  reject  $H_1$ . Otherwise accept  $H_1$ .

The fixed-sequence procedure controls the family-wise error rate in the strong sense because, for each null hypothesis, the testing is conditional upon rejecting all hypotheses earlier in the sequence (Dmitrienko, et al., 2009).

### 5.6.5. Multiple Comparison Adjustment for the Secondary Efficacy Endpoints

As type I error is only controlled for the primary, secondary endpoints will be considered exploratory. Each secondary endpoint will be tested independently and nominally following a hierarchical testing of doses like the one used for the primary. Interpretation of the analyses of secondary endpoints in the CSR should ensure to consider the dose ranging nature of the study.

### **5.6.6.** Examination of Subgroups

The following subgroups will be examined:

- 1. Current vs. ex-smokers
- 2. Chronic bronchitis vs. no chronic bronchitis at screening
- 3. Males vs. females.
- 4. Symptoms severity (MRC  $\leq$ 2 vs. MRC  $\geq$  2) at randomization
- 5. Age:  $(\ge 65 \text{ vs} < 65)$
- 6. Inhaled corticosteroid use versus no use (use of medications during the last 7 days of run-in phase).
- 7. By baseline FEV1 (> or <= 50% predicted)

Subgroup analyses will be performed for the primary and the selected secondary endpoints (see 5.4)

The MMRM model will be run on each subgroup separately.

### 6. Safety Endpoints

Safety measures that will be collected and investigated include adverse events (AEs), clinical




laboratory tests, vital signs, physical examination and electrocardiograms assessments (ECGs, 12-Lead and using 24 hour Holter monitors).

All safety analyses will be performed on the safety analysis set. Patients will be analyzed according to the treatment received. All safety summaries will present the five treatment groups.

### 6.1. Adverse Events

Treatment Emergent Adverse Events (TEAEs) are defined as all AEs which start after the first dose of study medication, or start prior to first dose of study medication and worsen, based on the investigator assessment of severity, on or after first dose of study medication.

Adverse events with completely missing onset dates will also be considered as treatment emergent. If any AE records contain only partial dates, these will be handled by imputation, as described in Section 3.8.4.

Table summaries will be produced summarizing AEs in the following ways:

- TEAEs
- TEAEs classified by maximum severity
- TEAEs classified with relationship to study medication
- TEAEs leading to study discontinuation
- Serious TEAEs
- Serious TEAEs classified by maximum severity
- Serious TEAEs classified with relationship to study medication
- Serious TEAEs leading to study discontinuation
- TEAEs with outcome death

### 6.1.1. Analysis of Adverse Events

Adverse events will be coded using MedDRA version 20 (June 2017).

All AE tables will be summarized by SOC and PT by treatment group, including the number of patients for each SOC and PT. Within each patient, multiple records of events mapping to a common MedDRA PT and SOC will be condensed into a single AE for incidence counts. Adverse Events will be reported by SOC and by PT in decreasing order of the highest active dose group of study medication (i.e 6.0 mg).

Listings of patients who discontinue the study for an AE, patients who experience an SAE and patients with AEs resulting in death will be presented.

### **6.2.** Clinical Laboratory Evaluations

- Change from baseline to Week 1 (Visit 3) in laboratory parameters
- Change from baseline to End of Study (Visit 6) in laboratory parameters

Laboratory parameters to be analyzed are:

- o Hematology: hemoglobin, hematocrit, total white cell count, leukocyte differential count and platelet count
- o Biochemistry: creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutamyl transferase, lactate dehydrogenase, creatine kinase, thyroid stimulating hormone, triiodothyronine and




thyroxine, glucose, potassium, sodium and calcium

o Urinalysis: leukocytes, blood, ketones, bilirubin, urobilinogen, protein and glucose.

### 6.2.1. Analysis of Clinical Laboratory Evaluation

Descriptive statistics (number of observations, mean, standard deviation, minimum, median and maximum values) for collected values and change from baseline will be summarized for clinical laboratory tests (hematology, biochemistry and urinalysis) at applicable visits, by treatment groups.

Selected laboratory test results will be classified by markedly abnormal criteria as normal or abnormal, according to Table 3 below. The number and percentage of patients with markedly abnormal laboratory results will be provided. No statistical testing will be performed on laboratory data.

| · | · - |
|---------------------------------|-----------------------------------|
| Parameter | Markedly Abnormally High Criteria |
| Alanine Amino Transferase (ALT) | >3 times Upper Limit of Normal |
| | Range |
| Alkaline Phosphatase | >3 times Upper Limit of Normal |
| | Range |
| Aspartate Amino Transferase | >3 times Upper Limit of Normal |
| (AST) | Range |
| Creatinine | 221 μmol/L |
| Gamma Glutamyl Transferase | >3 times Upper Limit of Normal |
| (GGT) | Range |
| Total Bilirubin | >3 times Upper Limit of Normal |
| | Range |

Table 3: Markedly abnormal ranges for clinical laboratory parameters

In addition, abnormal values (relative to the normal range) for hematology and biochemistry will be presented by treatment, patient, visit, and parameter in data listings (including all values of a parameter if at least one value was abnormal per patient). These listings will include: treatment, subject identifier, the laboratory parameter, units, visit number and study day, parameter value, an indicator for values outside of the reference range (H or L), the reference range, and an indicator for clinically significant out-of-range values.

All laboratory parameter results will be listed.

### 6.3. Electrocardiograms

- Change from baseline (pre-dose at Visit 2) to 2-hours post-dose at Day 1, Week 1, Week 2, Week 3 and End of study in ECG parameters
- Change from pre-dose to 2-hours post-dose at Week 1, Week 2, Week 3 and End of study in ECG parameters
- Clinically significant ECG abnormality during treatment period

ECG parameters to be analyzed are: QTcF Interval (msec), QRS Interval (msec), PR Interval (msec), RR (msec) and Heart rate (bpm).

### **6.3.1.** Analysis of ECG Evaluations

A 12-lead ECG will be recorded at Baseline and Screening, visits 2, 3, 4, 5 and end of study (or

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx




early termination). The overall ECG investigator interpretations will be summarized using a shift table comparing Baseline to time points. The ECG interpretations will be reported as "Normal", "Abnormal NCS (Not Clinically Significant)", or "Abnormal CS (Clinically Significant)". The denominators for the percentages will be the numbers of patients with ECG data at both the baseline and at the time point in question in each treatment group. The quantitative parameters listed in 6.3 will be summarized and listed.

### 6.3.2. Holter Monitors

• Change from screening to Week 4 in Holter parameters

The following parameter will be summarized:

Atrial Fibrillation Time in %, Supraventricular, Supraventricular Couplets, Supraventricular Runs, Ventricular Single, Ventricular Couplets, Ventricular Runs, Number of RR > 2 seconds The number of patients with Supraventricular or Ventricular runs, and the total number of runs will be also summarized at Screening and Week 4, presenting also the number of patients who had no runs at screening but had run at Week 4.

These parameters will also be listed together with the start and stop of Holter recording.

### 6.4. **Vital Signs**

- Change from baseline (pre-dose at Visit 2) to each post-dose assessment at Day 1, Week 1, Week 2, Week 3 and Week 4 in vital signs parameters
- Change from pre-dose to each post-dose assessment at Week 1, Week 2, Week 3 and Week 4 in vital signs parameters

Blood pressure (systolic and diastolic) and pulse rate will be measured at screening (visit 1) and pre-dose, 30 minutes and 1, 2, 4, 6, 8 and 12 hours post-dose at visits 2 and 6.

Blood pressure and pulse rate will be measured at pre-dose and 30 minutes, 1, 2 and 3 hours after dosing at visits 3 to 5.

### 6.4.1. Analysis of Vital Signs

Vital signs to be analyzed and presented are body weight, sitting blood pressure (systolic and diastolic), sitting pulse rate, and BMI. Vital signs at all study visits and changes from baseline at post-baseline visits will be summarized by visit for each treatment group using descriptive statistics.

Post-baseline results qualifying as Markedly Abnormal will be summarized by treatment group by parameter. Post-baseline markedly abnormal vital signs criteria are defined below:

Table 4: Markedly Abnormal Post-Baseline Vital Signs

| Vital Sign | Abnormally Low | Abnormally High |
|---|---|---|
| Parameter | | |
| Heart Rate (bpm) | A decrease from Baseline of | An increase from Baseline of |
| | ≥20 to a value ≤50 | ≥20 to a value ≥110 |
| Systolic blood | A decrease from Baseline of | An increase from Baseline of |
| pressure (mmHg) | ≥20 to a value ≤90 | ≥20 to a value ≥180 |
| Diastolic blood | A decrease from Baseline of | An increase from Baseline of |

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx




| pressure (mmHg) | ≥20 to a value ≤50 | ≥20 to a value ≥105 |
|------------------|--------------------|---------------------|
| Body weight (kg) | Loss of $\geq 5\%$ | Gain of $\geq 5\%$ |

Vital sign measurements will be presented by patient, visit and parameter in a data listing.

### 6.5. Physical Findings

The physical examination will be performed at screening and end of study (or early termination) and the results will only be listed.

### 6.6. Drug induced bronchospasm

Drug induced bronchospasm, defined as a decrease from pre-dose FEV<sub>1</sub> value of > 20% within the first hour after dosing.

### 6.6.1. Analysis of drug induced bronchospasm

The number of patients with at least one event of drug induced bronchospasm will be summarized by counts and percentage, overall and displayed by spirometry assessment (Day 1 and Week 1 to 4). The total number of events will also be displayed.

### 7. Pharmacokinetic

- Concentration of study medication at pre-dose assessment of Week 1 and Week 4
- Correlation of pre-dose concentration with trough FEV1 at Week 1 and at Week 4

### 7.1. Analysis of pharmacokinetic

The concentration of study medication will be summarized at week 1 and 4. The correlation with the pre-dose  $FEV_1$  value will be presented in a graphical representation. Pearson's correlation and its 95% CI will be presented as well.

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx



### 8. REFERENCES

- Decramer, M., Celli, B., Kesten, S., & al. (2009). Effect of tiotropium on outcomes in patients with moderate chronic obstructive pulmonary disease (UPLIFT): a prespecified subgroup analysis of a randomised controlled trial. *Lancet*, 1171-1178.
- Dmitrienko, A., Bretz, F., Westfall, P. H., Troendle, J., Wiens, B. L., Tamhane, A. C., & Hsu, J. C. (2009). Multiple testing methodology. Multiple Testing Problems in Pharmaceutical Statistics. *Chapman and Hall/CRC Press, New York*.
- Evidera. (2014). Retrieved from http://www.ema.europa.eu/docs/en\_GB/document\_library/Other/2015/04/WC50018544 3.pdf
- EXACT-PRO Initiative. (2014, October). *EMA*. Retrieved from http://www.ema.europa.eu/docs/en\_GB/document\_library/Other/2015/04/WC50018544 4.pdf
- Hajiro, T., Nishimura, K., Tsukino, M., Ikeda, A., Koyama, H., & Uzumi, T. (1998). Comparison of discriminative properties among disease-specific questionnaires for measuring health-related quality of life in patients with COPD. *American Journal of Respiratory and Critical Care Medicine*, 785-790.
- Jones, P. (2012, April). Retrieved from http://www.healthstatus.sgul.ac.uk/SGRQ\_download/sgrq-c-manual-april-2012.pdf
- Jones, P. W., Quirk, F. H., & Baveystock, C. M. (1991). The St George's Respiratory Questionnaire. *Respiratory Medicine*, 25-31.
- Mahler, D. A., & Wells, C. K. (1988). Evaluation of clinical methods for rating dyspnea. *Chest*, 580-586.
- Marcus, R., Peritz, E., & Gabriel, K. R. (1976). On Closed Testing Procedures With Special Reference to Ordered Analysis of Variance. *Biometrika*, 655-660.
- Maurer, W., Hothorn, L. A., & Lehmacher, W. (1995). Multiple Comparisons in Drug Clinical Trials and Preclinical Assays: A-priori ordered Hypotheses. *Testing Principles in Clinical and Preclinical Trials (J. Vollmar, editor) STuttgart, Gustav Fisher Verlag*, 3-18
- Meguro, M., Barley, E. A., Spencer, S., & Jones, P. W. (2007). Development and Validation of an Improved, COPD-Specific Version of the St. George Respiratory Questionnaire. *Chest*, 456-463.
- Miller, M. R., & al. (2005). Standardisation of spirometry. *European Respiratory Journal*, 153-161
- SAS Institute, Inc. (1999). SAS Procedures Guide, version 8. Cary, NC: SAS Institute.
- Siddiqui O, H. H. (2009). MMRM vs. LOCF: a comprehensive comparison based on simulation study and 25 NDA datasets. *Journal of biopharmaceutical statistics*, 19(2):227-46.
- Tamhane, A. C., & Logan, B. R. (2002). Multiple Test Procedures for Identifying the Minimum Effective and Maximum Safe Doses of a Drug. *Journal of the American Statistical Association*, 293-301.
- Westfall, P. H., & Krishen, A. (2001). Optimally weighted, fixed sequence, and gatekeeping multiple testing procedures. *Journal of Statistical Planning and Inference* 99, 25-40.
- WHO Collaborating Centre for International Drug Monitoring. (1993). *WHO Drug Dictionary*. Uppsala, Sweden (Box 26, S-751-03).



### Appendices 6

## Appendix 1: Schedule of Events 9.1.

| Visit | Visit 1a Screening<br>(Week-2 to -1) | Visit 1b<br>(Day after<br>Visit 1a) | Visit 2<br>Randomization | Visit 3 (Week 1<br>±1 day) | Visit 4 (Week 2<br>±1 day) | Visit 5<br>(Week 3 ±1<br>day) | Visit 6a<br>(Day<br>before<br>Visit 6b) | Visit 6b End of Study (Week 4 ±1 day or early termination) | Telephone<br>Follow-up (2<br>weeks after<br>Visit 6b ±3<br>days) |
|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | $X^{a}$ | | | | | | | | |
| Demographics, except body weight | X | | | | | | | | |
| Body weight | X | | | | | | | X | |
| Medical/surgical & disease history | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | X | | | | | | |
| Physical examination | X | | | | | | | X | |
| Nebulization inhalation training | | | X | | | | | | |
| Reversibility test | X | | | | | | | | |
| Randomization | | | X | | | | | | |
| Pregnancy test <sup>b</sup> | X | | X | X | X | X | | X | |
| Viral serology | X | | | | | | | | |
| Study medication inhalation | | | Xc | X | X | X | | X | |
| Spirometry | X | | $X^d$ | Xe | Xe | Xe | | $X^{d}$ | |
| Prior/concomitant medications | X | | X | X | X | X | | X | |
| Vital signs (blood pressure, pulse) | X | | Xf | Xg | Xs | Xg | | $X^{\mathrm{f}}$ | |

Version: 1.0 Version: 1.0 Version Date: 5<sup>th</sup> March 2018

### Verona Pharma RPL554-CO-203

# Statistical Analysis Plan

| s are now | |
|-------------|---|
| intiles are | 5 |
| Ith & Qui | 0 |
| IMS Health | |

| Visit | Visit 1a Screening<br>(Week-2 to -1) | Visit 1b<br>(Day after<br>Visit 1a) | Visit 2<br>Randomization | Visit 3 (Week 1<br>±1 day) | Visit 4 (Week 2<br>±1 day) | Visit 5<br>(Week 3 ±1<br>day) | Visit 6a<br>(Day<br>before<br>Visit 6b) | Visit 6b End<br>of Study<br>(Week 4 ±1<br>day or early<br>termination) | Telephone Follow-up (2 weeks after Visit 6b ±3 days) |
|---|---|---|---|---|---|---|---|---|---|
| ECG (QTcF and heart rate) | X | | Хh | Xh | Xh | Xh | | Xh | |
| Laboratory safety tests | X | | | × | | | | × | |
| Chest X-ray | X | | | | | | | | |
| Administer SGRQ-C,BDI/TDI and MRC breathlessness scale | | | įX | | Xi | | | Xi | |
| Administer PGAC questionnaire | | | | | X | | | X | |
| Dispense study medication and nebulizer | | | X | X | × | X | | | |
| Collect study medication and nebulizer | | | | X | × | × | | × | |
| Dispense compressor | | | X | | | | | | |
| Collect compressor | | | | | | | | X | |
| Dispense albuterol/salbutamol <sup>j</sup> | X | | | | | | | | |
| Trough PK blood sample | | | | X | | | | X | |
| Place Holter Monitor | X | | | | | | × | | |
| Remove Holter Monitor <sup>k</sup> | | X | | | | | | X | |
| Dispense symptom e-diary | X | | | | | | | | |

Version: 1.0 Version: 1.0 Version Date: 5<sup>th</sup> March 2018

# Statistical Analysis Plan



| Visit | Visit 1a Screening Visit 1b Visit (Week-2 to -1) (Day after Rand Visit 1a) | Visit 1b<br>(Day after<br>Visit 1a) | omization | 2 Visit 3 (Week 1 Visit 4 (Week 2 Visit ±1 day) ±1 day) (Weel day) = 4 day | Visit 4 (Week 2<br>±1 day) | × 3<br>⊞ | <u> </u> | 6a Visit 6b End Telephone of Study Follow-up (Week 4 ±1 weeks aff day or early Visit 6b : termination) days) | Telephone Follow-up (2 weeks after Visit 6b ±3 days) |
|---|---|---|---|---|---|---|---|---|---|
| Review symptom e-diary | | | X | X | X | X | | X | |
| Collect symptom e-diary | | | | | | | | X | |
| Adverse event questioning | X | | X | X | X | X | | X | X |
| Abhrevistime: BDI=Baseline Dyennes Index: ECG=electrocerdioorsm: ICS=inhaled conficosteroids: MRC=Medical Recearch Connocil: OToE=OT interval corrected using Fridericia's formula: | snnea Index. ECG=ele | etrocardioaram | · ICS=inhaled cortico | steroids: MRC=Medi | cal Pesearch Council | · OToE=OT inter | ual corrected in | eina Fridericia's | formula. |

Abbreviations: BDI=Baseline Dyspnea Index; ECG=electrocardiogram; ICS=inhaled corticosteroids; MRC=Medical Research Council; Q1cF=Q1 interval corrected using Fridericia's formula; PGAC=Patient Global Assessment of Change; PK=pharmacokinetics; SGRQ-C=St George's Respiratory Questionnaire-COPD specific; TDI=Transition Dyspnea Index

- Serum pregnancy test at Visit 1; urine pregnancy test at Visits 2-6 (a) Informed Consent may be obtained prior to screening visit
  (b) Serum pregnancy test at Visit 1: urine nreonancy test at Visit 1.
- At Visit 2, study medication is to be administered at the study clinic twice; first, just after randomization and again 12 hours later once all assessments are complete © ©
  - Spirometry at Visits 2 and 6 is performed 15 minutes pre-dose, followed by 30 minutes and 1, 2, 3, 4, 6, 8 and 12 hours post-dose
- Spirometry at Visits 3, 4, and 5 are performed 15 minutes pre-dose, followed by 30 minutes and 1, 2, and 3 hours post-dose
  - Vital signs at Visits 2 and 6 are measured pre-dose and 30 minutes, 1, 2, 4, 6, 8, and 12 hours post-dose
    - Vital signs at Visits 3, 4, and 5 are measured pre-dose and 30 minutes, 1, 2 and 3 hours post-dose
- ECG at Visits 2 through 6 is performed pre-dose and 2 hours post-dose
  - BDI administered at Visit 2, TDI administered at Visits 4 and 6
- A second canister of albuterol/salbutamol may be dispensed during the study if necessary
  - Holter is to be removed 24 hours ( $\pm$  1 hour) after placement

Version: 1.0

Version Date: 5th March 2018



### 9.2. Appendix 2: EXACT-PRO and E-RS Scoring Instructions

The following instructions are from the user manual for EXACT-PRO, version 7.0 (EXACT-PRO Initiative, 2014)

- Raw scores are assigned to each item response option as shown in Table 7 below. Please note that items 3, 8, 9, 10, 11 and 14 have separate scoring instructions, namely with the same raw score being assigned to several answer options.
- Sum the item-level raw scores of the 14 EXACT items to form the raw summed score
- For each raw summed score, look up the corresponding EXACT Total score from Table 6 below.

### Notes:

- 1. EXACT total scores range from 0 to 100
- 2. If the EXACT total score is 0, set to missing.
- 3. The Evaluating Respiratory Symptoms (E-RS) part of the <u>EXACT tool consists</u> of the first 11 items, broken down as follows (Evidera, 2014):
  - a. RS-Breathlessness: items 7, 8, 9, 10 and 11 (score range: 0-17);
  - b. RS-Cough & Sputum: items 2, 3 and 4 (score range: 0-11);
  - c. RS-Chest Symptoms: items 1, 5 and 6 (score range: 0-12).

### Scoring the domains:

The following respiratory domains are included in the EXACT measure: Breathlessness, Cough/Sputum and Chest Symptoms.

Items are assigned to specific domains as follows (please note that items 4, 12, 13 and 14 do not correspond to a domain and hence, are not used in domain-specific analyses):

- Breathlessness: items 7, 8, 9, 10 and 11
- Cough and Sputum: items 2 and 3
- Chest Symptoms: items 1, 5 and 6

### Score the domains as follows:


- For each day, sum the item-level raw scores of the items comprising the domain to form the domain raw summed score. If no diary entry exists for a given day, leave the domain raw summed score missing.
- For each domain raw summed score, look up the corresponding EXACT domain score from Table 7
- If no diary entry exists for a given day, leave the EXACT domain score missing.
- If the daily EXACT domain score is 0, set it to missing.

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx Author: Eleonora Chiossi



Table 5: Annotated EXACT for raw score assignment

| Table 5: Annotated EXACT for raw score assignment | T |
|---|---|
| 1. Did your chest feel congested today? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 2. How often did you cough today? | 0.Not at all |
| | 1.Rarely |
| | 2.Occasionally |
| | 3.Frequently |
| | 4.Almost constantly |
| 3. How much mucus (phlegm) did you bring up when | 0.None at all |
| coughing today? | 1.A little |
| | 1.Some |
| | 2.A great deal |
| | 3.A very great deal |
| 4. How difficult was it to bring up mucus (phlegm) | 0.Not at all |
| today? | 1.Slightly |
| 10 440) | 2.Moderately |
| | 3.Quite a bit |
| | 4.Extremely |
| 5. Did you have chest discomfort today? | 0.Not at all |
| 3. Did you have eliest discomfort today: | 1.Slight |
| | 2.Moderate |
| | 3.Severe |
| | 4.Extreme |
| 6. Did your chest feel tight today? | 0.Not at all |
| o. Did your chest reer tight today: | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 7. Were you breathless today? | 0.Not at all |
| 7. Were you oreamess today: | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 8.Describe how breathless you were today | 0.Unaware of breathlessness |
| 8.Describe now breatmess you were today | 1.Breathless during strenuous |
| | activity strendous |
| | 2.Breathless during light activity |
| | 4.5 |
| | 3.Breathless when washing or dressing |
| | 3.Present when resting |
| 0. Ware you short of breath today when performing your | 0.Not at all |
| 9. Were you short of breath today when performing your usual personal care activities like washing or dressing? | |
| usual personal care activities like washing of dressing? | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 4.Too breathless to do these |

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx Author: Eleonora Chiossi



| 10. Were you short of breath today when performing your | 0.Not at all |
|---|---|
| usual indoor activities like cleaning or household work? | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 3.Too breathless to do these |
| 11. Were you short of breath today when performing your | 0.Not at all |
| usual activities outside the home such as yard work or | 1.Slightly |
| errands? | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 3.Too breathless to do these |
| 12. Were you tired or weak today? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 13. Last night, was your sleep disturbed? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 14. How scared or worried were you about your lung | 0.Not at all |
| problems today? | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |

Version: 1.0  Version Date: 5<sup>th</sup> March 2018



Table 6: Raw Summed Score to Scale Conversion Table for EXACT Total Score

| Raw Summed | EXACT Total | | EXACT Total |
|------------|-------------|-------|-------------|
| Score | Score | Score | Score |
| 0 | 0 | 26 | 50 |
| 1 | 8 | 27 | 51 |
| 2 | 13 | 28 | 52 |
| 3 | 17 | 29 | 53 |
| 4 | 20 | 30 | 54 |
| 5 | 23 | 31 | 55 |
| 6 | 25 | 32 | 57 |
| 7 | 27 | 33 | 58 |
| 8 | 28 | 34 | 59 |
| 9 | 30 | 35 | 60 |
| 10 | 31 | 36 | 61 |
| 11 | 33 | 37 | 63 |
| 12 | 34 | 38 | 64 |
| 13 | 36 | 39 | 65 |
| 14 | 37 | 40 | 67 |
| 15 | 38 | 41 | 68 |
| 16 | 39 | 42 | 70 |
| 17 | 40 | 43 | 72 |
| 18 | 41 | 44 | 73 |
| 19 | 42 | 45 | 75 |
| 20 | 43 | 46 | 77 |
| 21 | 44 | 47 | 80 |
| 22 | 46 | 48 | 83 |
| 23 | 47 | 49 | 87 |
| 24 | 48 | 50 | 92 |
| 25 | 49 | 51 | 100 |

Version: 1.0  Version Date: 5<sup>th</sup> March 2018



Table 7: Raw Summed Score to Scale Score Conversion Table for EXACT Domains

| Domain Raw | Breathlessness | Cough & Sputum | <b>Chest Symptoms</b> |
|---|---|---|---|
| <b>Summed Score</b> | <b>Domain Score</b> | <b>Domain Score</b> | <b>Domain Score</b> |
| 0 | 0 | 0 | 0 |
| 1 | 11 | 13 | 12 |
| 2 | 19 | 25 | 23 |
| 3 | 25 | 39 | 31 |
| 4 | 30 | 56 | 38 |
| 5 | 34 | 72 | 45 |
| 6 | 38 | 86 | 52 |
| 7 | 42 | 100 | 58 |
| 8 | 45 | | 65 |
| 9 | 48 | | 72 |
| 10 | 52 | | 79 |
| 11 | 56 | | 88 |
| 12 | 60 | | 100 |
| 13 | 65 | | |
| 14 | 71 | | |
| 15 | 78 | | |
| 16 | 87 | | |
| 17 | 100 | | |



### 9.3. Appendix 3: SGRQ-C

**Table 9: SGRQ-C Item weights** 

| Table 9: SGRQ-C Item weights Question | Aneware | Weight |
|---|---|---|
| Part 1 | Answers | weignt |
| Question 1: I cough | | 1 |
| Question 1. I cough | Most days | 80.6 |
| | | 46.3 |
| | Several days With chest infections | 28.1 |
| Overtice 2. I being your able one (construe) | Not at all | 0.0 |
| Question 2: I bring up phlegm (sputum) | Most dove | 76.8 |
| | Most days | 47.0 |
| | Several days With chest infections | 30.2 |
| O | Not at all | 0.0 |
| Question 3: I have shortness of breath | Mark Jana | 97.2 |
| | Most days | 87.2 |
| | Several days | 50.3 |
| Overtion 4. There etterly forthere: | Not at all | 0.0 |
| Question 4: I have attacks of wheezing | Mont done | 96.2 |
| | Most days | 86.2 |
| | Several days | 71.0 |
| | A few days | 45.6 |
| | With chest infections | 36.4 |
| 0 5 5 11 | Not at all | 0.0 |
| Question 5: How many attacks of chest | | 00.1 |
| trouble have you had | 3 or more | 80.1 |
| | 1 or 2 attacks | 52.3 |
| | None | 0.0 |
| Question 6: How often do you have good | | 02.2 |
| days (with little chest trouble) | None | 93.3 |
| | A few | 76.6 |
| | Most are good | 38.5 |
| | Every day | 0.0 |
| Question 7: If you have a wheeze, is it | | |
| worse in the morning? | No | 0.0 |
| | Yes | 62.0 |
| Part 2 | | |
| Question 8: How would you describe your | | |
| chest condition? | The most important problem I have | 82.9 |
| | Causes me a few problems | 34.6 |
| | Causes no problem | 0.0 |
| Question 9: Questions about what | | |
| activities usually make you feel breathless | Getting washed or dressed | 82.8 |
| | Walking around the home | 80.2 |
| | Walking outside on the level | 81.4 |
| | Walking up a flight of stairs | 76.1 |
| | Walking up hills | 75.1 |
| Question 10: More questions about your | | |
| cough and breathlessness | My cough hurts | 81.1 |

Document:U:\My documents\ad hoc\Mark\Final SAP\Verona RPL554-CO-203 SAP v1.0.docx Author: Eleonora Chiossi



| - | My cough makes me tired | 79.1 |
|---|---|---|
| | I get breathless when I talk | 84.5 |
| | I get breathless when I bend over | 76.8 |
| | My cough or breathing disturbs my | 87.9 |
| | sleep | 01.7 |
| | I get exhausted easily | 84.0 |
| Question 11: Questions about other effects | I get exhausted easily | 04.0 |
| your chest trouble may have on you | | |
| Jour 611600 1100010 11111 1111 11 11 11 11 11 11 | My cough or breathing is embarrassing in public | 74.1 |
| | My chest trouble is a nuisance to my family, friends or neighbors | 79.1 |
| | I get afraid or panic when I cannot get my breath | 87.7 |
| | I feel that I am not in control of my chest problem | 90.1 |
| | I have become frail or an invalid because of my chest | 89.9 |
| | Exercise is not safe for me | 75.7 |
| | Everything seems too much of an effort | 84.5 |
| Question 12: Questions about how | | |
| activities may be affected by your breathing | I take a long time to get washed or dressed | 74.2 |
| | I cannot take a bath or shower, or I take a long time | 81.0 |
| | I walk more slowly than other people, or I stop for rests | 71.7 |
| | Jobs such as housework take a long time, or I have to stop for rests | 70.6 |
| | If I walk up one flight of stairs, I have to go slowly or stop | 71.6 |
| | If I hurry or walk fast, I have to stop or slow down | 72.3 |
| | My breathing makes it difficult to do things such as walk up hills, carry things up stairs, light gardening such as weeding, dance, play bowls or play golf | 74.5 |
| | My breathing makes it difficult to do things such as carry heavy loads, dig the garden or shovel snow, jog or walk at 5 miles per hour, play tennis or swim | 71.4 |
| Question 13: We would like to know how | | |
| your chest trouble actually affects your | I cannot play sports or games | 64.8 |
| daily life | I cannot go out for entertainment or recreation | 79.8 |
| | I cannot go out of the house to do the shopping | 81.0 |



| | I cannot do housework | 79.1 |
|---|---|---|
| | I cannot move far from my bed or | 94.0 |
| | chair | |
| Question 14: Tick the statement which you | | |
| think best describes how your chest affects | It does not stop me doing anything I | 0.0 |
| you | would like to do | |
| | It stops me doing one or two things I | 42.0 |
| | would like to do | |
| | It stops me doing most of the things I | 84.2 |
| | would like to do | |
| | It stops me doing everything I would | 96.7 |
| | like to do | |

### 9.4. Appendix 4: SAS code for efficacy analysis

```
proc mixed data=efficacy;
class subject trt country visit;
model outcome= trt visit trt*visit b_fev /ddfm=kr;
repeated visit/ sub=subject type=un;
lsmeans trt*visit/ cl diff;
```

### run;

where outcome is the change from baseline

 $Document: U:\My\ documents\ad\ hoc\Mark\Final\ SAP\Verona\ RPL554-CO-203\ SAP\ v1.0.docx\ Author:\ Eleonora\ Chiossi$ 

Version: 1.0  Version Date: 5<sup>th</sup> March 2018